CLINICAL TRIAL: NCT03959046
Title: Giving Information Strategically and Transparently in Hematopoietic Stem Cell Transplantation/Bone Marrow Transplantation
Brief Title: GIST in Hematopoietic Stem Cell Transplantation/Bone Marrow Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been withdrawn due to delays caused by COVID-19 and practical barriers to conducting the study.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1807019470; 5R35CA197730 (NIH)
Record Dates: First submitted 2019-05-14; First posted 2019-05-22 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2021-06

CONDITIONS: Liquid Tumor; Cancer; Psychological Feedback
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patient participants will be seeing the same physician they usually see, and they won't know if their physician was assigned to GIST or not.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GIST (Experimental): GIST is an alternative way of speaking to patients. In order for patients to get the "gist," Hematologists will ensure that patients walk away from their initial consultation understanding: why they are candidates for bone marrow transplant (BMT), what the process for BMT is, and the major risks involved.
  Interventions: Behavioral: GIST
- Usual Care (No Intervention): These are physician and patient participants that will communicate in their normal, unchanged way.

INTERVENTIONS:
Behavioral: GIST — The GIST intervention will train physicians in an alternative way of communicating with their patients.
  Arms: GIST

SUMMARY:
The purpose of this study is to assess the efficacy of using GIST language when speaking to patients about bone marrow and hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Hematopoietic stem cell/bone marrow transplantation (HSCT/BMT) is a high-risk, complicated procedure that is poorly understood by patients, posing a challenge for informed decision-making. One study found that 69.7% of patients needed more information about HSCT to make an informed decision. Furthermore, for most patients who seek HSCT/BMT as treatment, transplantation is the only viable option for long-term, disease-free survival. In light of limited options, it is often assumed that patients will choose to undergo transplantation by default, which might undermine efforts to ensure that patients are fully informed. Given the context in which the decision to undergo transplantation are made, there is a clear and present need to ensure that patients are properly informed about HSCT/BMT.

Unfortunately, this need does not seem to be adequately met. For example, studies have shown that patients tend not to remember rates of risks and complications. One study found that after completing HSCT, patients recalled a mortality risk rate lower than those provided by physicians at their initial consultation (20% vs. 30%, respectively). Findings such as this highlight the need to improve the informed consent process for patients confronting the decision to undergo HSCT/BMT.

The present study aims to improve the informed consent process by proposing a new approach to patient-physician communication, called Giving Information Simply and Transparently (GIST), that will train physicians to speak more understandably, with the goal of improving patients understanding of the procedures they intend to pursue. This approach is based upon Dr. Valerie Reyna's Fuzzy Trace Theory which posits that patients focus on the bottom-line gist of information when formulating their treatment preferences. Patient understanding will be tested via assessments administered after their consultation visit, 30 days after initiation of chemotherapy, and 100 days after initiation of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* acute myeloid leukemia with high or intermediate risk in first complete remission acute myeloid leukemia OR myelodysplastic syndrome beyond first remission chronic myeloid leukemia with accelerated phase or blast crisis acute lymphocytic leukemia Myeloma lymphoma with a sensitive relapse lymphoma with a resistant relapse first time undergoing consultation at this institution's HSCT/BMT program Fluent in English

Exclusion Criteria:

* Cognitively impaired
* Not fluent in English

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change from 1 week post baseline understanding at 3 months | 1 week, 1 month and 3 months from baseline (T2, T3, and T4)
  Evidence that patients assigned to physicians trained in the GIST approach will have improved recall of information and be able to answer more questions correctly about HSCT/BMT than those assigned to care as usual. The researchers have developed a brief assessment of patient knowledge of: a) why the participants are a candidate for HSCT/BMT; b) what the procedure involves; c) risks and benefits posed by HSCT/BMT. The assessment will consist of multiple choice questions, with one fill-in-the-diagram question. The high score is 90, and the low score is 18. A score of 90 means that the participant fully understands the three points listed above. A score of 18 means that the participant has little to no understanding of the three points listed above.

SECONDARY OUTCOMES:
Patient's emotional acceptance of their illness | 1 week, 1 month and 3 months from baseline (T2, T3, and T4)
  We will use 5 relevant items from the validated PEACE scale which asks patients about how accepting they are of their illness. Responses include "not at all", "to a slight extent", "to some extent", "to a large extent". The questionnaire is composed of two combined subscales: a 2-item "Peaceful Acceptance" and a 3-item "Struggle with Illness" subscale. Both subscales are associated with patients' self-reported peacefulness "Struggle with Illness" scores are associated with acknowledgement of cognitive terminal illness. The low score for this scale is 5 (indicating little acceptance) and the high score is 20 (indicating high acceptance).
Patient's emotional acceptance of their lives | 1 week, 1 month and 3 months from baseline (T2, T3, and T4)
  The MEPSI is an 8 item questionnaire (shortened from the original) that asks patients to respond to phrases regarding how they view their lives. Responses include "not at all", "to a slight extent", "to some extent", "to a large extent". The questionnaire is composed of two combined subscales: a 4 item "Positive" subscale and a 4-item "Negative" subscale. The low score for this scale is 8 (indicating little acceptance) and the high score is 32 (indicating high acceptance).

OTHER OUTCOMES:
The Human Connection (THC) Scale | One week, one month and three months from baseline (T2, T3, and T4)
  The effect on changing physician communication on patient-physician relationships will be measured by The Human Connection (THC) scale. THC is a validated 16 item questionnaire that measures the extent to which patients felt a sense of mutual understanding, caring, and trust with their physicians. Patients are asked to circle one of four phrases that answers the questions. The 16-item THC questionnaire was internally consistent (Cronbach's α =.90) and valid, based on its expected positive association with emotional acceptance of the terminal illness (r=.31, P<.0001). Scores range from 16 (the lowest score, indicating a weak therapeutic alliance) and 64 (the high score, indicating a strong therapeutic alliance).
Levels of anxiety and depression in patients | 1 week, 1 month and 3 months from baseline (T2, T3, and T4)
  levels of anxiety and depression will be assessed via the Hospital Anxiety and Depression Scale (HADS). It is a verified and brief 14-item tool that asks patients to choose a 1 out of 4 possible responses to each statement, with each response being assigned to a score of 0, 1, 2, or 3. 7 statements correspond to measuring depression, while the other 7 corresponding to measuring anxiety. Score of 0-7 indicates that the patient is "normal; 8-10 indicates the patient is borderline; and 11-21 indicates abnormal.
Health Literacy in older adults compared to younger adults | Baseline, 1 week, 1 month and 3 months from baseline (T1, T2, T3, and T4)
  The researchers have developed a brief assessment of patient knowledge of: a) why the participants are a candidate for HSCT/BMT; b) what the procedure involves; c) risks and benefits posed by HSCT/BMT. The assessment will consist of multiple choice questions, with one fill-in-the-diagram question. The high score is 90, and the low score is 18. A score of 90 means that the participant fully understands the three points listed above. A score of 18 means that the participant has little to no understanding of the three points listed above. We will compare the scores of older adults (>65) to younger adults (<65) to see which group overall has a higher score.
Assessment of patient's health literacy | 1 week, 1 month and 3 months from baseline (T2, T3, and T4)
  Assessment of patient's health literacy via Rapid Estimate of Adult Literacy in Medicine - Short Form(REALM-SF) will be administered to control for variable health literacy. REALM-SF is a validated and brief literacy assessment tool of a patient's health literacy. REALM-SF consists of a list of 7 medically related words that is shown to the patient. Patients are asked to read the words out loud in order of the list, with the option of saying "pass" when they encounter a word that they do not recognize, allowing them to move onto the next word; alternatively, patients taking longer than 5 seconds to read a word will be told to move onto the next word by the interviewer. Each word a patient recognizes is a point that is used to score the assessment. 0 points is equivalent to a 3rd grade reading level, 1-3 points is equivalent to a 4th to 6th grade level, 4-6 points is equivalent to a 7th to 8th grade level, and 7 points is equivalent to at least a high school level.

CONTACTS AND LOCATIONS:
Overall Officials: Holly G Prigerson, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). Results will be presented at scientific meetings in the form of posters and oral presentations
Time Frame: Data will be available after the final analysis is completed. No end date.
Access Criteria: Upon request, we will provide the dataset to qualified investigators under a Data Use Agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.